



Study Number:

Participant Identification Number for this trial:

## **CONSENT FORM**

Title of Project: Colo-Pro Pilot: A pilot randomised controlled single blind trial to compare standard single dose antibiotic prophylaxis to antibiotic prophylaxis administered as a bolus-continuous infusion for the prevention of surgical site infections in adults undergoing colorectal surgery.

Name of Researcher: Andrew Kirby

| Name of Person taking consent | | Date | S | Signature | | |
|---|---|---|---|---|---|---|
| Name of Participant | | Date | <br>S | ignature | | |
| 6. | I agree to take part in | the above study. | | | | |
| 5. | <ol> <li>I agree to a rectal swab being collected before my operation, and blood samples to be<br/>collected during my operation.</li> </ol> | | | | | |
| 4. | I understand that the information collected about me will be used to support other research in the future, and may be shared anonymously with other researchers. | | | | | |
| 3. | I understand that relevant sections of my medical notes and data collected during the study, may be looked at by individuals from Leeds Teaching Hospitals or regulatory authorities, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | | | | | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | | | | | |
| 1. | I confirm that I have read the information sheet dated (version) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | | | | | |
| INAIII | e of Researcher: Andr | ew Kirby | | | Pleas | e initial box |